CLINICAL TRIAL: NCT03098784
Title: Nanoparticles Emitted by Aircraft Engines, Impact on Respiratory Function
Acronym: NPAF
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Aix Marseille Université (Other); LBM- Nanosecurity platform - CEA Grenoble (Unknown); LR2N - Nanosecurity platform - CEA Grenoble (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8755; 2011-A00646-35 (Other: RCB number)
Record Dates: First submitted 2016-08-23; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Function
Keywords: airport environment; Air France; flightline employees; administrative employees
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Air France employees working near runways: Air France personnel mainly working in physical proximity to the runways of the Marseille Marignane or Parisian airports.
  Intervention: Exposure to aircraft exhaust
  Interventions: Other: Exposure to aircraft exhaust
- Air France employees working inside: Air France personnel working mainly inside buildings at the Marseille Marignane or Parisian airports.
  Intervention: Non exposure to aircraft exhaust
  Interventions: Other: Non exposure to aircraft exhaust

INTERVENTIONS:
Other: Exposure to aircraft exhaust — The exposed group is made up of Air France personnel mainly working in physical proximity to the runways of the Marseille Marignane or Parisian airports. These people are subject to direct exposure to exhaust from aircraft engines.
  Groups: Air France employees working near runways
Other: Non exposure to aircraft exhaust — The non-exposed group is made up of Air France personnel working mainly inside buildings at the Marseille Marignane or Parisian airports. These people are not subject to direct exposure to exhaust from aircraft engines.
  Groups: Air France employees working inside

SUMMARY:
The goal of this study is to assess the respiratory health of the Air France company's employees working in the Marseilles and Paris airports (flight line and administrative employees). This study was promoted by the Montpellier CHRU, Regional University Hospital Centre (ANSM identification number 2011-A00646-35). It allowes voluntary employees to be involved. They answer a lifestyle survey and perform a spirometry, an exhaled CO measurement and a sampling of exhaled air condensate (EAC). A metrological study of particles emitted by aircraft engines and found in the airport environment will be conducted and the elementary chemical composition analysis, as well a sieve analysis of particles present in the EAC will be conducted.

DETAILED DESCRIPTION:
Air traffic is increasing, raising concern about local pollution and its adverse health effects on the people living in the vicinity of large airports. However, the highest risk is probably occupational exposure due to proximity. Jet exhaust is one of the main concerns at an airport and may have a health impact, particularly on the respiratory tract. Current studies are neither numerous enough nor strong enough to prove this kind of association. Yet, more and more people work in airports, and occupational exposure to jet exhaust is a fact. In 1999, the effect of occupational exposure to aircraft fuel and jet exhaust on pulmonary function and respiratory symptoms in Birmingham International Airport (Birmingham, UK) workers was reported. This work suggested that there was a link between high occupational exposure to aviation fuel or jet exhaust and excess respiratory tract symptoms, consistent with the presence of a respiratory irritant. It was a cross-sectional survey using a questionnaire filled out by the participants themselves. Respiratory and immunological function assessments and an exhaled carbon monoxide measurement were conducted with male full-time airport workers classified into three groups according to their exposure level.

The study will be presented to the volunteering subjects during an occupational medical appointment concerning their company. The information letter will be provided as well as the informed consent form to be filled for the study. Once the subjects have agreed to participate, self-surveys on their lifestyle habits will be filled and EACand urine samplings will be taken during one same consultation, in addition to exhaled CO and No measurements. This consultation will also include a spirometry test. The employees' workstation data will be collected. Therefore, the volunteers' participation is limited to one single visit including non-invasive examinations and self-surveys.

Method details:

* Survey: The survey breaks down into 2 parts, with a total of 94 items. The first part bears on the employees' respiratory health condition, essentially grounded on the validated EGEA survey. The rest focuses on employees' lifestyle habits, both professionally (outdoor and indoor working time, trade, type of exposure, etc.) and personally (geographical situation of the home, type of town or community, heating system, usual mode of cooking, etc.). The survey is anonymised and the answers are automatically read by datascan process.
* Spirometry: This method allows a non-invasive, simple and repeatable assessment of the respiratory function. It is indispensable to clearly explain the process to the patient. The patient sits with his or her back straight during the process. Once the subject and the device are ready, the subject deeply breathes in to fill the lungs then fully expires into the spirometer. Then the subject breathes in fully and forcedly in order to obtain the inspiratory curve. The spirometry results are compared with theoretical or predicted values determined based on patient's age, gender, size and ethnic group. Consequently, according to the subject's breathing speed and force intensity, measurements of vital capacity (VC) or forced vital capacity (FVC) are obtained. The curves will allow the other variables to be deduced, such as maximum expiratory volume per second (MEVS) or peak expiratory flow (PEF), or mean expiratory flows (MEF 25-75).
* Exhaled CO measurement (confounding factors of the respiratory function, in order to reflect the smoking status):the employee blows into the device's single-use cardboard mouthpiece after a deep inspiration followed by a fifteen-second apnea computed by the device. The measurement in part per million (ppm) is immediately displayed on the device to quantify the severity of CO intoxication. This measurement is simple and repeatable.
* Exhaled air condensate:for EAC acquisition. In fact, the RTube device is well adapted to non-invasion collection on the companies' sites. It will be used according to the recommendations from the American Thoracic Society and the EuropeanRespiratory Society. The R tube will be pre-treated as in the first study (intensive washing in order to abate background noise) and "white" R tubeswill be collected all through the study to check the method's detection limit. Briefly, the collection with nose blocked lasts for 15 minutes during which the subject breathes normally through the device. The mouth is rinsed with water before collection and the subject is asked to refrain from drinking or eating during the previous hour. This will allow ca. 1.4 ml to be collected (mean EACvolume collected during the first study over a 15-minute breathing time).
* Metrology:as this is a recent subject, there is no consensus so far on the most representative unit of measurement for employee exposure. Similarly, no current device allows all parameters to be obtained:quantitative data (particle content/cm3, sieve distribution, developed surface area of the alveolar fraction likely to be exposed in the breathing apparatus) and qualitative data (morphology, aggregation/agglomeration status, listof constitutive chemical elements). These experts' surveys require the implementation of different equipment. The method is based on personal metrology, use of portable and individual systems, as well as fixed installation metrology, organised into a single sampling by means of a cane to which the various measuring instruments are connected (Condensation ParticleCounter, ElectrostaticLow Pressure Impactor, Scanning MobilityParticleSizer, FastMobilityParticleSizer, Nanometer Surface Area Monitor, Alveolar Sensor, Alveolar Inhalable Thoracic sensor).An independent counter (Condensation ParticleCounter) allows background evolution to be monitored. Membrane sensors (such as the Giliansampling pump with membrane support) will also complement the process. They will be used as portable systems, on the employees involved in the study. Finally, the samples will be analysed by means of a SEM (Scanning Electron Microscope),model 5500 from Hitachi, associated with an energy-dispersive EDX system (X analysis system - Noranmodel from the Thermocompany).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be given free and informed consent and signed the consent
* Subject must be affiliated or beneficiary in a health insurance plan

Exclusion Criteria:

* Subject has a cons-indication (or an incompatible combination therapy) for the realization of the EFR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Air France employees working in the Marseilles or Parisian airports (flightline and administrative employees)
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The quantity of nanoparticules present in exhaled air condensate | 1 day (Day of inclusion (D0)
  The quantity of nanoparticules present in exhaled air condensate

SECONDARY OUTCOMES:
Exhaled CO measurement | 1 day (Day of inclusion (D0)
  Exhaled CO measurement
Exhaled NO measurement | 1 day (Day of inclusion (D0)
  Exhaled NO measurement
Exhaled air condensate | 1 day (Day of inclusion (D0)
  Exhaled air condensate
oxidative stress marker (8 isoprostane) | 1 day (Day of inclusion (D0)
  oxidative stress marker (8 isoprostane)
plasma mass spectrometry which allows the simultaneous assaying of 17 elements | 1 day (Day of inclusion (D0)
  plasma mass spectrometry which allows the simultaneous assaying of 17 elements (Zn, Al, Ti, Co, Cu, Zr, Ni, Cr, Ga, In, Mn, Fe, Se, Cd, Ge, Be)
Lung function | 1 day (Day of inclusion (D0)
  Spirometry value

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS MOLINARI, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
NC